CLINICAL TRIAL: NCT07081724
Title: Opt In - Implementation and Evaluation of an Early Intervention Program for Children Waiting to Receive an Autism Diagnosis
Brief Title: "Opt-In" Early Intervention Program for Children Waiting to Receive an Autism Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2401010296A003; 1R01HD114761-01A1 (NIH)
Record Dates: First submitted 2025-06-27; First posted 2025-07-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Autism
Keywords: randomized controlled trial; autism early intervention
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: post-intervention outcomes will be assessed by clinicians who will be blind to group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPT-IN intervention (Experimental): Participants randomized to the experimental condition will be given access to the the "Online Parent Training in Early Behavioral Intervention" (OPT-In-Early; Dai et al., 2018, 2021,2022), a self-directed online resource for caregivers of children with autism or high likelihood of autism. The OPT-In-Early program includes 14 modules (6 mandatory, 8 optional) comprising text and video demonstrations to teach caregivers effective methods for improving their children's language, social, and adaptive skills (e.g., using utensils, toilet training), and reducing their children's disruptive behavior. Parents in the OPT-In-Early condition will be also offered the option to schedule brief support calls with a clinician for the duration of the 6-month trial, with a limit of three calls per week. These optional support calls are designed to provide parents with clarification and guidance on how to navigate the website materials, including selection of the appropriate modules.
  Interventions: Behavioral: Online Parent Training in Early Behavioral Intervention (OPT-In-Early)
- Waitlist (No Intervention): Child-parent dyads randomly assigned to the waitlist group will not receive immediate access to the OPT-In intervention or any other intervention. However, after 6 month (equivalent to the the 6-month intervention period) they will be given access to the OPT-In intervention. However, outcomes will not be measured for these participants.

INTERVENTIONS:
Behavioral: Online Parent Training in Early Behavioral Intervention (OPT-In-Early) — the "Online Parent Training in Early Behavioral Intervention" (OPT-In-Early; Dai et al., 2018, 2021,2022) is a self-directed online resource for caregivers of children with autism or high likelihood of autism. The OPT-In-Early program includes 14 modules (6 mandatory, 8 optional) comprising text and video demonstrations to teach caregivers effective methods for improving their children's language, social, and adaptive skills (e.g., using utensils, toilet training), and reducing their children's disruptive behavior. Parents are taught how to facilitate joint attention, imitation, pretend play, language, sharing, emotional engagement, social play, and self-help skills such as feeding and dressing in their child using behavioral principles (e.g. prompting, shaping and fading) during play and naturalistic daily routines. The optional modules cover such topics as picky eating and toilet training.
  Arms: OPT-IN intervention

SUMMARY:
A growing body of literature documents the benefits of parent-mediated interventions for autism starting early in life . However, the median age of diagnosis in the US continues to be 49 months. Even following formal diagnosis, services often do not begin for another 9 months on average. Such harmful delays in accessing autism-specific early interventions are potentially avoidable, as caregivers of children later diagnosed with autism identify concerns about their child's development by 13 months on average - including difficulties that can be successfully addressed through evidence-based intervention practices. Wait times to receive a formal diagnosis of autism are such a significant barrier that they have been referred to as a "crisis" in the field, with parents reporting an average wait time of 1.2 years in the US. The current proposal focuses on circumventing the roadblock of delayed access to diagnosis and intervention by empowering caregivers to address their children's needs before a diagnosis is established.

This will be accomplished through the implementation and evaluation of the "Online Parent Training in Early Behavioral Intervention (OPT-In-Early)", a self-directed online resource for caregivers of autistic children which will be made available during their enrollment in waitlists for a diagnostic evaluation. Key features of OPT-In-Early include: (a) a comprehensive scope (i.e., multiple developmental domains are addressed), (b) a focus on evidence-based Naturalistic Developmental Behavioral Intervention strategies, (c) a combination of required and optional modules, so that caregivers can focus on areas most relevant to their child's needs, and (d) access to online materials designed for self-directed implementation, as well as access to remote consultation with a clinician for advice, clarification and support (including on selection of appropriate modules).

Following an alternative approach to the current "parental concerns - then enrollment in waitlist - then clinical diagnosis - then intervention", the program is designed to counteract the harmful and frustrating inaction that characterizes the waitlist time with timely action designed to address areas of concern that caregivers have already identified and should be empowered to address. This has the potential to capitalize on the window of opportunity of early brain plasticity, thus maximizing outcomes, and to reduce the anxiety associated with the lack of services that characterizes the period of "passive waiting" for a formal diagnosis. To evaluate the utility of this innovative resource, the following specific aims will be addressed:

1. Comparing outcomes for 120 toddlers aged 16-48 months whose caregivers are on a waitlist to receive a formal autism diagnosis, randomly assigned to receive either OPT-In-Early or no intervention during a six-month period. The investigators predict that (a) children randomized to the OPT-In-Early condition will have superior gains as reflected in the Goal Attainment Scaling, changes in adaptive behavior and social communication standardized measures, and (b) their families will experience superior improvements in their well-being.
2. Examining implementation outcomes of feasibility and acceptability of the intervention. The investigators predict high acceptability and feasibility for the OPT-In-Early content and format, as indicated by end-users' responses to standardized measures reflecting 80%+ agreement on the feasibility and acceptability of the program.
3. As an exploratory aim, investigators will examine theoretically- and empirically- motivated factors associated with intervention uptake and child outcomes, including demographic profiles and child clinical presentation.

Examining whether accessing and using OPT-In-Early during waitlist time is a viable alternative to the current "first diagnosis then intervention" format (for all children, or for children with specific profiles and needs) is a critical step toward promoting a more efficient intervention delivery model, bridging the gap between onset of parental concerns and availability of intervention practices designed to target such concerns.

DETAILED DESCRIPTION:
BACKGROUND. The increasing prevalence of autism spectrum disorder (ASD), now at 1 in 36 children, highlights an urgent need for early interventions that are both effective and efficient, given the social and economic impact of the challenges experienced by individuals on the autism spectrum and their families. Several clinical trials have documented the benefits of parent-mediated interventions starting early in life, even before a formal autism diagnosis is established. Symptoms of autism manifest across the lifespan and can be diagnosed as early as 12 months of age. Although parents often identify concerns about their child's development during the first two years of life, the median age of diagnosis in the United States continues to be 49 months. Even following formal diagnosis, services often do not begin for another 9 months. These cumulative waiting times often result in children receiving minimal early intervention prior to school entry. Additionally, health disparities disproportionally affect access to services for families from minoritized and socioeconomically disadvantaged backgrounds. Families who are low-income, have low parental educational attainment, or are from minoritized racial and ethnic backgrounds not only experience delays in receiving diagnoses, but are also less likely to receive high-quality services following diagnosis. These inequities have been exacerbated by the COVID-19 pandemic.

Barriers to accessing diagnostic services limit the opportunity to receive autism-specific interventions at the age for which they are shown to be maximally beneficial. Children on the autism spectrum whose needs are not addressed in a timely fashion are at an increased risk of impairments in cognitive, adaptive, and social dimensions of well-being, as well as physical and mental health issues. Further, the 'passive waiting' time in the waitlist is harmful for parental wellbeing and mental health, with research reporting feelings of frustration, worry, and stress in parents experiencing the yearlong 'odyssey' from initial concerns to diagnosis and intervention referral.

Importantly, such harmful delays in accessing autism-specific early interventions are potentially avoidable, as many caregivers of children later diagnosed with autism identify concerns about their child's development before her or his second birthday, often as early as 13 months of age. Many difficulties identified by parents during infancy and toddlerhood can be successfully addressed through evidence-based intervention practices. For example, early emerging differences in verbal and nonverbal communication are amenable to improvements through targeted parent-mediated interventions, with benefits documented across multiple dimensions of wellbeing (i.e., adaptive and social-communicative functioning).

Despite advances in this area, the potential benefits of early interventions remain largely untapped, as wait times to receive a formal diagnosis of autism are such a significant barrier that they have been referred to as a "crisis" in the field, with parents reporting an average wait time of 1.2 years in the US. The American Academy of Pediatrics recommends simultaneous referrals for clinical diagnostic evaluation and early intervention for young children with suspected autism - however, most children without an autism diagnosis receive low-intensity, generic early interventions rather than autism-specific early intervention programs that rely on evidence-based practices. Accordingly, key stakeholders, including caregivers and providers, have voiced the need for facilitating earlier access to intervention options to counteract the harmful impact of the waitlist crisis. Accordingly, the current project focuses on circumventing the roadblock of delayed access to diagnosis and intervention by empowering caregivers to address their children's needs while they are waiting to be seen for a formal diagnosis.

One viable option to accomplish this goal is the delivery of parent-mediated intervention programs that do not require a previous diagnosis or enrollment in formal early intervention services. In particular, recent research has shown the promise of self-directed online intervention programs for caregivers of autistic children. These programs involve independent access to online resources that caregivers can utilize at their own pace and individualize to their own children by selecting content relevant to the specific difficulties experienced by their children. Implementation of the intervention strategies might be exclusively self-directed (i.e., parents deliver the intervention strategy without any assistance from a provider) or based on a hybrid format, whereby a clinician is available to provide guidance and clarification related to the program's content, although without explicit coaching and feedback. Across formats, self-directed programs do not rely on diagnostic and intervention services for eligibility, insurance and billing purposes, providing a potential avenue for circumventing the roadblock of delayed access to diagnosis and intervention. Research has documented that despite not being coached by experienced clinicians, caregivers have expressed a high degree of acceptability and satisfaction with the self-directed format, demonstrated fidelity of implementation, experienced gains in knowledge and their use of the intervention strategies was associated with child improvements following parent completion of programs. However, substantial variation in outcomes in response to different self-directed programs was documented, and existing research only focuses on children who were already diagnosed. Therefore, the potential impact of a self-directed intervention program during families' enrolment in waitlists for a diagnostic evaluation remains unexplored.

Against this background, our project focuses the implementation and evaluation of the "Online Parent Training in Early Behavioral Intervention" (OPT-In-Early), a self-directed online resource for caregivers of children with autism or high likelihood of autism which will be made available during their enrolment in waitlists for a diagnostic evaluation. Key features of Opt-In-Early include: (a) a comprehensive scope (i.e., multiple domains are addressed), (b) the use of a Naturalistic Developmental Behavioral Intervention approach, i.e., evidence-supported strategies that blend behavioral and developmental components to address the needs of autistic children and their families, (c) a combination of required and optional modules, so that caregivers can learn autism-specific strategies and focus on areas most relevant to their specific child's needs, and (d) a hybrid format including access to web-based materials designed for self-directed implementation, as well as optional access to remote consultation with a clinician for advice, clarification and support (e.g., selection of appropriate modules).

APPROACH.

The overarching goal of our project is to evaluate the utility of the OPT-In-Early program for caregivers of toddlers who are on a waitlist for receiving diagnostic services. The OPT-In-Early program centers on the use of naturalistic, developmental, and behavioral principles to increase motivation and engagement, teach skills, and generalize skills across settings. The program emphasizes the importance of utilizing the parent-child relationship, the child's interests, and daily routines to facilitate skill acquisition, and to create developmentally appropriate learning experiences, to value small gains, and to use evidence-based applied behavior analytic principles including task analysis, prompting and prompt fading, and contingent reinforcement. Optional modules focus on specific needs, such as toilet training and picky eating. To evaluate whether the OPT-In-Early program is an acceptable and effective tool for caregivers who are on a waitlist for receiving diagnostic services, the following specific aims will be addressed:

1. Comparing outcomes for 120 toddlers aged 16-48 months whose caregivers are on a waitlist to receive a formal autism diagnosis, randomly assigned to receive either OPT-In-Early or no intervention for six months period. The investigators hypothesize that children randomized to the OPT-In-Early condition will have superior gains.
2. Examining feasibility and acceptability of the intervention (both hypothesized to be high).
3. As an exploratory aim, the investigators will examine theoretically- and empirically- motivated factors associated with intervention engagement and child outcomes.

Participants and Setting. Participants will be 120 toddler-caregiver dyads (with each dyad including one toddler and one caregiver) who are on a waitlist to receive a formal diagnostic evaluation due to autism concerns identified by either parents or professionals. As the study does not involve in-person contact between investigators and participants, participants will be recruited across any geographical area.

Inclusion criteria include (a) age between 16-48 months, (b) parental consent, (c) being on a waitlist to receive a formal diagnostic evaluation at the time of parent consent due to autism concerns, (d) parents speak English, (e) an initial score of 8 or greater or Follow-Up score of 2 or greater on the Modified Checklist for Autism in Toddlers, Revised, with Follow-Up (M-CHAT-R/F) as an indication of autism likelihood.

Exclusion criteria include (a) having already received a formal diagnosis of autism, (b) enrolment in early intervention programs delivering more than 5 h per week of evidence-based autism-specific interventions at the time of consent, (c) child has a gestational age less than 36 weeks associated with a birth weight less than 2500 g, (d) the child is not yet walking, or has severe hearing and/or vision impairment that is uncorrected with aids, or known neurological disorder or genetic syndrome (e.g., Down syndrome).

Research Design. Our aims will be addressed using an intent-to-treat randomized controlled trial, with participants randomized to either the OPT-In-Early intervention or a waitlist control condition, stratified by age, language level and parental education. Data will be collected from each family prior to random assignment (baseline) and following completion of the 6-month trial period (or earlier for families electing to discontinuing their participation from the trial). The investigators will use REDCap, a HIPAA-compliant data management software to store data. To ensure data accuracy, data will be doubled entered by independent research team members, when not collected directly via REDCap.

Study flow. The study flow is articulated in the 5 steps. In step 1 participants will be recruited through our extensive network of hospitals and clinical centers who provide diagnostic evaluations for autism, who will show study flyers in their waiting rooms and websites and inform families enrolled in their waitlist about the opportunity to participate. Interested caregivers will complete a phone screen to learn more about the study and to confirm eligibility.

In step 2 caregivers who are invited and consented to the RCT will complete baseline assessments prior to randomization through an online procedure that includes completing online forms and phone interviews conducted by a clinician blind to group allocation and study hypotheses. Assessment measures will include standardized measures indexing broad adaptive functioning and severity of autism symptoms, as well as an idiographic measure capturing goals specific for each dyad. During the baseline assessment, a detailed description of the specific goals that each participant family wants to achieve with their child (e.g., addressing difficulties with verbal communication, toilet training, food refusal) will be obtained using Goal Attainment Scaling procedures. As part of the process, parents will be also asked to provide 3 to 5 "baseline goal" videos of 5- to 20-min in length illustrating the current level of performance in the skill that they are planning to address (one video for each goal) - such as, for example, a video illustrating lack of responsiveness to the child's name being called, a second video illustrating food refusal during lunch, and a third video illustrating the child having a tantrum when asked to brush her teeth. The study coordinator will provide guidance on the videos (e.g., duration, camera angle) to ensure consistency across participants. These videos will be used for later coding of change occurring from baseline to post-intervention.

In step 3 each child-parent dyad will be randomly assigned to either the OPT-In-Early condition or the waitlist condition using the online randomization program randomize.net. Randomization will be concealed from clinicians assessing outcomes and stratified by child age (older than vs. equal to or younger than 24 months) language level (expressive language age equivalence score on the Vineland older than vs. equal to or younger than 18 months, reflecting benchmarks of pre-verbal vs. verbal functioning) and parental education (dichotomized as "some college or less" vs "bachelor's degree or more"), based on the literature suggesting that these factors are associated with response to early intervention.

In step 4, child-parent dyads randomly assigned to the OPT-In-Early condition will be granted access to the online password-protected OPT-In-Early website for up to 6 months, and provided guidance on the selection of modules within OPT-In-Early that are relevant to the goals caregivers indicated as their priorities during the baseline assessment. The OPT-In-Early program includes 14 modules (6 mandatory, 8 optional) comprising text and video demonstrations to teach caregivers effective methods for improving their children's language, social, and adaptive skills (e.g., using utensils, toilet training), and reducing their children's disruptive behavior. Parents are taught how to facilitate joint attention, imitation, pretend play, language, sharing, emotional engagement, social play, and self-help skills such as feeding and dressing in their child using behavioral principles (e.g. prompting, shaping and fading) during play and naturalistic daily routines. The optional modules cover such topics as picky eating and toilet training. Parents in the OPT-In-Early condition will be also offered the option to schedule brief (i.e.,15-30 min) support calls with a clinician with a BCBA credential and expertise in each module's content (e.g., PECS, behavior assessment) for the duration of the 6-month trial, with a limit of three calls per week. These optional support calls are designed to provide parents with clarification and guidance on how to navigate the website materials, including selection of the appropriate modules. However, no instruction or feedback on how the parents are implementing the strategies (i.e., fidelity monitoring) will be provided, consistent with the self-directed nature of the intervention.

Child-parent dyads randomly assigned to the waitlist group will receive access to the OPT-In-Early website immediately after their second (i.e., "post-intervention") assessment. Therefore, all participants will be given access to the intervention, with the only difference being that access will be given after a 6-month wait time for dyads assigned to the waitlist group (although intervention outcomes will not be assessed for those assigned to the waitlist group after receiving OPT-In).

In step 5, post-intervention outcomes will be assessed by clinicians who will be blind to group assignment after 6 months from the baseline assessments. A group comparison approach was favored over a cross-over design due to the risk of carry-over effects. The post- intervention evaluation will include the same measures administered at baseline.

MEASURES The Modified Checklist for Autism in Toddlers, Revised with Follow-Up (M-CHAT-R/F) is a 20-item (yes/no) parent-report, autism-specific screener; although initially validated for ages 16-30m, evidence supports use to 48 m. The M-CHAT-R/F provides scores that are indicative of "low likelihood" (< 3), "high likelihood" (≥8), or "moderate likelihood" (3-7) for autism. Moderate likelihood scores trigger the structured Follow-Up questions, with two at-risk items on the follow-up signaling the need for evaluation referral. Initial M-CHAT-R items requires 5 min to complete and follow-up questions require an additional 10 min. The M-CHAT-R/F will be used to determine eligibility, based on the presence of clinical concerns operationalized as an initial score of 8 or greater or follow-up score of 2 or greater, and to quantify the degree of clinical concerns at baseline. The M-CHAT-R/F will be also used to characterize participants at baseline and will not be repeated at post-intervention as it is not used as an outcome measure.

The Goal Attainment Scaling (GAS) will be used as a proximal measure of intervention response, i.e., a measure that captures changes in the specific goals selected for each participant. The GAS is designed to assess an individual's progress on a goal in relation to their baseline performance, and has been successfully utilized to capture proximal response to interventions for individuals on the autism spectrum, particularly for interventions that include different targets for different participants. Stakeholders have increasingly endorsed measurement of goals relevant to the needs of specific individuals within the autism population. Additionally, the GAS was selected to account for the heterogeneity of intervention targets within the OPT-In-Early intervention, whereby selection of modules and targets differ across participants. The GAS includes standardized procedures to generate a common metric of intervention change across participants who have different intervention goals, as articulated below.

GAS Baseline assessment and goal setting. For each participant, goals will be developed based on detailed information obtained in a parent interview at the baseline assessment. Each goal is designed to identify an area in which the child is experiencing difficulties (e.g., picky eating, toilet training, self-injurious behavior) that caregivers want to address by teaching specific skills. Caregivers will be encouraged to identify three to five goals that are priorities for their family. The number of goals will vary across participants but is not expected to differ across groups, as goals will be established prior to randomization - however the number of goals targeted for each participant will be considered in the statistical analyses. The stringent standardization criteria detailed in Ruble et al., 2012 will be used to ensure that the goals are unambiguously operationalized and measurable based on: (1) the description of the skill planned to be targeted, (2) the prompt level required by the child for engaging in the targeted skill, and (3) the criterion for success. Caregivers will be asked to provide a set of 5- to 20-min videos (one for each to-be-targeted skill) illustrating their child's current level of performance in the skills that they are planning to target.

GAS post-intervention outcome assessment. At the post intervention evaluation, caregivers will be asked to provide a second set of videos, one for each targeted goal, capturing their child's behavior in relation to the same situations/behaviors videotaped at baseline, so that change in relation to the specific goals identified by caregivers can be examined.

GAS video collection procedures. For both phases of video collection, caregivers will be provided guidance by study personnel and asked to provide videos that capture the average or typical performance/ behavior currently displayed by their child with reference to the target goal, rather than the child's 'best' behavior. Previous research has shown that intervention participants typically do not use unrepresentative behavior samples in their selections of videos to be submitted for coding of goal attainment. Given the heterogeneity of needs in this population, the investigators expect different caregivers to identify different goals important to them, and to select different OPT-In-Early modules accordingly (e.g., the 'picky eating' module for a child displaying severe food refusal, or the 'toilet training' module for a child experiencing challenges in that domain). Consistent with the idiographic nature of the Goal Attainment Scaling, this will result in specific content and different quantity of videos from each participant.

GAS rating. Following previous research, videos will be rated according to the GAS standard procedures whereby goals at baseline are assigned a score of -2 and are then scored on a 5-point scale at post-treatment with positive changes in score from baseline indicating increasingly positive benchmarks of improvement from the baseline to post-intervention. Consistent with previous trials that have used the GAS as an outcome measure, a trained clinician blind to study group and hypotheses will complete the ratings. A coding manual will be developed following Ruble et al., and 20% of videos will be coded by a senior rater (co-I de Marchena) to establish interrater reliability. Participant GAS scores will be averaged across modules to derive an overall score of goal attainment.

The following measures will be used as secondary distal outcome measures .

The Vineland Scales of Adaptive Behavior-3 (VABS-3), a standardized measure of adaptive functioning, will be administered to all participants at pre- and post-treatment to evaluate change occurring in adaptive behavior across groups. Previous research has documented that this measure has robust psychometric properties, is sensitive to change in response to early intervention, and captures dimensions that are highly valued by stakeholders.

Participants' caregivers will also complete the Parenting Stress Index-4, Short-Form (PSI), a standardized measure of parental wellbeing with robust psychometric properties, which has been used in previous research with a similar population. The PSI will be completed at baseline and post-intervention to quantify intervention-related changes in stress. A focus on parenting stress has been endorsed as a top priority by autistic advocates as well as caregivers.

The Autism Impact Measure (AIM) is a caregiver-report questionnaire that focuses on the frequency and impact of autism-associated challenges in social interaction, communication, peer interaction as well as repetitive and unusual behaviors. It will be administered at baseline and post-intervention to assess changes in social and communication functioning across groups. The AIM has been shown to have robust psychometric properties.

The following measures will be administered to measure intervention feasibility and acceptability. Caregivers of participants randomized to the OPT-In condition will be administered the Acceptability of Intervention Measure and the Feasibility of Intervention Measure. These two standardized measures assess the extent to which end-users believe the intervention was acceptable and could be successfully carried out. To gain insight on feasibility and acceptability issues related to specific modules, participants will be asked to rate the program overall as well as each specific module they utilized. Both scales demonstrated robust discriminant validity and reliability.

From onset of intervention until completion of post-intervention evaluation, caregivers will complete a monthly update either electronically or by phone (based on their preferences). Caregivers across conditions will report details about all interventions, services and supports the child is receiving outside the OPT-In-Early program. In addition, caregivers will be asked about any new medical conditions, medical updates, and updates on diagnostic evaluations. These factors will be accounted for in our analyses of the OPT-In-Early program.

Finally, Opt-In-Early website usage analytics, including the frequency of access and the specific modules being accessed will be used to provide a measure of the caregivers' engagement with the website content. This information, together with a detailed log on the frequency of optional support calls by participants, will be used to examine the link between usage of the available resources and outcomes.

ANALYTIC APPROACH Power analysis. The primary aim is to compare changes in the GAS rating in the OPT-In-Early intervention group to changes in the waitlist group from baseline to after 6 months. Although no research to our knowledge has used the GAS for this population, previous studies that have used the GAS to measure intervention-related change in children on the autism spectrum documented an improvement of 2.1 GAS units with a standard deviation of 0.79. Given our study population and goals, the investigators calculated the sample sizes required to detect change in GAS rating ranging from 0.5 to 2. The power table calculations are based on a mixed-model analysis with 2 observations per participant (e.g., baseline and 6 months). For example, to detect a difference in change in GAS rating in the OPT-In group compared to the waitlist group of 1.0, 76 participants (38 per group) are needed to achieve 80% power with a standard deviation of 1.0, within-subject correlation of 0.01, and significance level (alpha) of 0.025. Given the possibility of 30% dropout, a conservative enrollment plan of 120 participants (60 per group) will be implemented to ensure detection of a minimum difference of 1.0 in GAS rating.

Statistical Plan. The investigators will employ best practices for collecting, verifying, managing, and analyzing data. Data will be examined to identify outliers, batch effects, and significant departures from normality for continuous outcomes. Accuracy and explanation for any identified outliers will be explored and dealt with accordingly. Analyses will be performed with and without extreme scores to evaluate their influence on the results. As some attrition is inevitable, baseline data also will be used to assess for non-equivalent attrition between groups and to subsequently support statistically controlling for any bias in attrition. This is consistent with our goal of conducting intent-to-treat analyses for all specific and exploratory aims discussed below.

Aim 1 - Primary outcome. The investigators will employ a linear mixed effects modeling approach to compare change (baseline to 6 months) in GAS rating in the OPT-In-Early group to change in the waitlist group. The model will include participant-level random intercepts. Fixed effects in the model will include time (baseline, 6 months), treatment group, and the interaction between time and treatment group. Our model will include age, language level (as measured via the Vineland), M-CHAT-R/F score (as an indicator of clinical severity at baseline), and parental education as fixed effects. Given the RCT study design, the investigators expect balance at baseline on most covariates. However, the investigators will examine balance on other relevant variables - including family size, and other interventions received during the trial - and consider their inclusion in the model accordingly. Using this model, the investigators will estimate mean and 95% confidence intervals for GAS rating at baseline and 6 months. From these means, the investigators will estimate the change in GAS rating in the OPT-In-Early group and the waitlist group. Next, the investigators will contrast those changes with one another to quantify the intervention effect.

Secondary distal outcomes. To investigate differences in VABS-3, PSI-4 and AIM score, the investigators will use a similar statistical approach to the one outlined for the primary proximal outcome. Mixed effects models will be used to estimate and contrast outcome changes in the OPT-In-Early group to changes in the waitlist group.

Aim 2 - Feasibility and acceptability of the OPT-In-Early content and format will be investigated using the Acceptability of Intervention Measure and Feasibility of Intervention Measure, which use a 5-point Likert scale ranging from 1 (completely disagree) to 5 (completely agree). The investigators will classify participant agreement on feasibility and acceptability using as "in agreement" (average response score of ≥ 4) or "not in agreement" (average response score < 4). Responses will be summarized using counts and percentages. The investigators will test whether at least 80% of participants are in agreement on each metric using one-sample tests of proportion.

Aim 3 - In an exploratory analysis, the investigators will investigate theoretically and empirically motivated factors that may affect intervention engagement and child outcomes. Exploratory outcomes: engagement. Engagement outcomes will include engagement with program content (frequency of module access) and use of support calls (frequency of calls), evaluated separately. Explanatory variables of interest (i.e. putative predictors) will include diagnosis during participation in the trial, chronological age, baseline adaptive behavior and social communication functioning, and demographic factors (including parental education, employment status and family size). The investigators will model the relationship between these explanatory variables and rate of each of the outcomes using Poisson regression models. These models will be used to estimate and contrast the average rate of module access or rate of support calls by predictor group. Exploratory outcomes: child change. The investigators will examine whether putative predictors including program engagement (frequency of module access and frequency of calls), baseline adaptive behavior and social communication, chronological age, M-CHAT-R/F score, presence/absence of a diagnosis of autism during the trial, other interventions received during the trial, and demographic factors will affect change in GAS rating, assessed using a mixed effects modeling approach based on the approach described for Aim 1 (substituting the predictor variables for treatment group).

Examining whether accessing and using OPT-In-Early during waitlist time is a viable alternative to the current "first diagnosis then intervention" format (for all children, or for children with specific profiles and needs) can be a critical step toward promoting a more efficient delivery model intervention, bridging the gap between timing of parental concerns and availability of intervention practices designed to target such concerns.

ELIGIBILITY:
Inclusion Criteria:

* age between 16-48 months,
* parental consent
* being on a waitlist to receive a formal diagnostic evaluation at the time of parent consent due to autism concerns
* parents speak English
* an initial score of 8 or greater or Follow-Up score of 2 or greater on the Modified Checklist for Autism in Toddlers, Revised, with Follow-Up (M-CHAT-R/F; Robins et al., 2014) as an indication of autism likelihood.

Exclusion Criteria:

* having already received a formal diagnosis of autism
* enrollment in early intervention programs delivering more than 5 h per week of evidence-based autism-specific interventions at the time of consent
* child has a gestational age less than 36 weeks associated with a birth weight less than 2500 g
* the child is not yet walking, or has severe hearing and/or vision impairment that is uncorrected with aids, or known neurological disorder or genetic syndrome (e.g., Down syndrome).

Ages: 16 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling | Within 30 days from consent
  The Goal Attainment Scaling (GAS) is a proximal measure of intervention response, i.e., a measure that captures changes in the specific goals selected for each participant. The GAS is designed to assess an individual's progress on a goal in relation to their baseline performance. The GAS includes standardized procedures to generate a common metric of intervention change across participants who have different intervention goals. For each participant, goals are developed based on areas in which the child is experiencing difficulties (e.g., picky eating, toilet training, self-injurious behavior) that caregivers want to address by teaching specific skills. Videos provided by the caregivers at pre- and post- intervention are rated according to the GAS standard procedures on a 5-point scale, whereby positive changes in score from baseline indicating increasingly positive benchmarks of improvement from the baseline to post-intervention.

SECONDARY OUTCOMES:
Vineland Scales of Adaptive Behavior-3 | Within 30 days from consent
  The Vineland Scales of Adaptive Behavior-3 (VABS-3), a standardized parent interview measuring adaptive functioning, will be administered to all participants at pre- and post-treatment to evaluate change occurring in adaptive behavior across groups. Previous research has documented that this measure has robust psychometric properties, is sensitive to change in response to early intervention, and captures dimensions that are highly valued by stakeholders. Higher scores in the VABS indicate more advanced adaptive skills.
Parenting Stress Index-4, Short-Form | Within 30 days from consent
  The Parenting Stress Index-4, Short-Form (PSI), a standardized measure of parental wellbeing with robust psychometric properties, which has been used in previous research with a similar population. Higher scores in the PSI indicate more parenting stress.
Autism Impact Measure (AIM) | Within 30 days from consent
  The Autism Impact Measure (AIM) is a caregiver-report questionnaire that focuses on the frequency and impact of autism-associated challenges in social interaction, communication, peer interaction as well as repetitive and unusual behaviors. It will be administered at baseline and post-intervention to assess changes in social and communication functioning across groups. The AIM has been shown to have robust psychometric properties. Higher scores in the AIM indicate higher frequency and impact of autism-associated challenges.

OTHER OUTCOMES:
Acceptability of Intervention Measure | Within 14 days of intervention completion (approximately 6 months from intervention start)
  The Acceptability of Intervention Measure is a standardized measure assessing the extent to which end-users believe the intervention was acceptable. Participants are asked to rate the acceptability of the program overall as well as each specific module they utilized. Higher scores indicate higher acceptability.
Feasibility of Intervention Measure | Within 14 days of intervention completion within 14 days of intervention completion (approximately 6 months from intervention start)
  The Feasibility of Intervention Measure is a standardized questionnaire assessing the extent to which end-users believe the intervention can be successfully carried out. To gain insight on feasibility issues related to specific modules, participants will be asked to rate the program overall as well as each specific module they utilized. Higher scores indicate higher feasibility.

CONTACTS AND LOCATIONS:
Locations (1):
- A.J. Drexel Autism Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in the primary publication will be shared, including demographic information, outcome measures, and adverse events.
  The data will be made available beginning 6 months after publication of the primary results and will be available for 3 years thereafter.
  Researchers who provide a methodologically sound proposal and have appropriate institutional review board (IRB) approval will be granted access. Requests will be reviewed by the study's PI.

REFERENCES:
- [Background] Ruble L, McGrew JH, Toland MD. Goal attainment scaling as an outcome measure in randomized controlled trials of psychosocial interventions in autism. J Autism Dev Disord. 2012 Sep;42(9):1974-83. doi: 10.1007/s10803-012-1446-7. PMID 22271197